CLINICAL TRIAL: NCT05773001
Title: Macrophage Regulation of Ozone-Induced Lung Inflammation
Acronym: MOLI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Tighe, MD (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor-Investigator, Robert Tighe, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Pro00110603; 1R01ES034350-01 (NIH)
Record Dates: First submitted 2023-03-03; First posted 2023-03-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: SARS-CoV-2 Pneumonia
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Other): No history of SARS-CoV-2
  Interventions: Drug: Ozone
- Cohort 2 (Other): Documented mild SARS-CoV-2 infection
  Interventions: Drug: Ozone
- Cohort 3 (Other): SARS-CoV-2 pneumonia
  Interventions: Drug: Ozone

INTERVENTIONS:
Drug: Ozone — Subjects will perform alternating 15 minutes rest with 15 minutes treadmill walk exercise periods for 135 minutes in while breathing Ozone (O3).
  Other Names: O3

SUMMARY:
The purpose of this research study to understand how prior respiratory infections affect the susceptibility to lung inflammation following environmental exposures.

DETAILED DESCRIPTION:
Study participants will undergo a 1-day screening that includes a blood draw and breathing testing, return for a two-day series of testing to include blood draw, and brief breathing test before and after an inhaled challenge with either filtered air (FA) or ozone (O3). Participants return the next day for a brief breathing test, a blood draw and a procedure called bronchoscopy to evaluate the lung after the challenge.

Participants then return 18 - 20 days later to repeat the two-day series of testing to be challenged with the exposure not received on the first series, (FA or O3). Each visit will take about 3 - 3.5 hours. Follow-up phone calls from the study team will occur at 24 hours after each 2-day test series.

Total study duration is about one to one-and a half months.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18-55 yrs. of age (No subject will be excluded from the study on the basis of gender or ethnicity)
* Individuals with knowledge of prior SARS-CoV-2 infection history allowing them to be segregated into one of three cohorts

  * Cohort 1 - No history of SARS-CoV-2 infection (defined as no symptoms consisted with SARS-CoV-2 nor history of a positive SARS-CoV-2 test)
  * Cohort 2 - Documented mild SARS-CoV-2 infection (a positive test, either PCR- or antigen-based) but with mild to no symptoms and no evidence of a lower respiratory tract infection (including no hospitalization, and no oxygen use)
  * Cohort 3 - History of SARS-CoV-2 infection and symptoms/imaging consistent with a lower respiratory tract infection who have recovered, are >6 months out from their infection, and have normal lung function (spirometry with FVC, FEV1 and FEV1/FVC)

    * There will be no maximal period from SARS-CoV-2 infection for inclusion in the study, the minimal period will be >6 months out from infection

Exclusion Criteria:

* Individuals with prior SARS-CoV-2 pneumonia who have ongoing respiratory symptoms, are still using supplemental oxygen, or have abnormal lung function
* Individuals with prior SARS-CoV-2 infection that cannot provide documentation of a positive test
* Current smokers of tobacco products including e-cigarettes or those with previous smoking history within the prior 5 years
* Pregnant women and women who are presently lactating.
* Subjects that have received antibiotic administration or an upper respiratory infection within the previous 4 weeks
* College and graduate students or employees who are under direct supervision by any of the investigators in this protocol
* Alcohol or illicit substance abuse
* Chronic cardio/pulmonary respiratory disorders or other medical conditions as determined by the investigator
* Increased airway hyperresponsiveness at baseline as measured by a positive methacholine challenge response (methacholine PC20 FEV1 < 4 mg/ml)
* Subjects will be requested to refrain from antihistamines, nonsteroidal anti-inflammatory agents, antioxidants (e.g. beta-carotene, selenium, and lutein) and supplemental vitamins (e.g. C and E), for 1 week prior to, and during testing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in the abundance of monocyte-derived alveolar macrophages | Baseline, Day 18-20
  - Change in the abundance of monocyte-derived alveolar macrophages and association to measures of O3-induced inflammation (BAL cell neutrophils, albumin and cytokine production)

SECONDARY OUTCOMES:
Change in the abundance of autonomous CSF-1 expression in alveolar macrophages | Baseline, Day 18-20
  - Change in the abundance of autonomous CSF-1 expression in alveolar macrophages and association to measures of O3-induced inflammation
Association between prior evidence of COVID pneumonia | Baseline, Day 18-20
  Association between prior evidence of COVID pneumonia, when compared to non-COVID infected individuals, and O3-induced inflammation
Association between prior evidence of COVID infection without pneumonia | Baseline, Day 18-20
  Association between prior evidence of COVID infection without pneumonia, when compared to non-COVID infected individuals and O3-induced inflammation

OTHER OUTCOMES:
Change in composition of BAL immune cells following O3 exposure | Baseline, Day 18-20
  Change in composition of BAL immune cells following O3 exposure will identify unique immune cells driving inflammation and physiologic responses
Comparison between BAL immune cells and immune cells obtained from bronchial brushings | Baseline, Day 18-20
  Comparison between BAL immune cells and immune cells obtained from bronchial brushings and the relationship to O3 induced inflammation and physiologic responses
Interactions between airway epithelial cells and immune cells | Baseline, Day 18-20
  o Interactions between airway epithelial cells and immune cells by RNA-sequencing to define an "interactome"

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tighe, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No